CLINICAL TRIAL: NCT03961139
Title: Continuous Versus Intermittent Bolus Feeding in Very Preterm Infants - Effects on Respiratory Morbidity: A Multicentre Randomised Controlled Clinical Trial
Brief Title: Continuous Versus Intermittent Bolus Feeding in Very Preterm Infants - Effect on Respiratory Morbidity
Acronym: CONFER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018/00773
Record Dates: First submitted 2019-05-15; First posted 2019-05-23 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-05

CONDITIONS: Chronic Lung Disease of Prematurity; Bronchopulmonary Dysplasia
Keywords: Prematurity; Randomised control trial (RCT); BPD; CLD; continuous feeding
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Intervention Model Description: Randomised-controlled trial with 2 parallel groups (1:1 ratio). Control group: intermittent bolus intra-gastric tube feeding (BF), Intervention group: continuous intra-gastric tube feeding (CF). Not blinded.
  Stratified randomization along following birth weight groups:
  1. </=750 g
  2. 751 - 1000 g
  3. 1001 -1250 g Method of randomisation: Computer generated randomization codes stored in sealed opaque envelopes.
  Intervention started by 72 hours of life (more than trophic feed volume achieved) and continued until an infant reaches a weight of 1.6 kg and is determined by the attending Neonatologist to be ready to commence oral feeding by breast or bottle, or when an infant attains a post-conceptional age of 36 weeks, whichever is earlier.
  Continuous fed is delivered through a nasogastric tube by a syringe pump over 3hrs with 1 hour of break - 6 cycles a day. Feed volume, type of feed, feed increment regulated by the clinical team.
  Intention to treat analysis.
Masking Description: na. Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous feeding (CF) (Experimental): Infants fed through a naso or orogastric tube in a continuous fashion using syringe pump. Each feed cycle is of 4 hours (3 hrs continuous feeding and 1 hour rest). 6 feed cycles in a day.
  Feed volume increment per day is as per departmental protocol and same as comparator arm.
  Interventions: Other: Method of feeding; continuous feeding OR bolus feeding
- Bolus feeding (BF) (Active Comparator): Infants fed through a naso or orogastric tube in a gravity dependent bolus feeding every 2-3 hours. Each feed would take approximately 10 minutes.
  Feed volume increment per day is as per departmental protocol and same as experimental arm.
  Interventions: Other: Method of feeding; continuous feeding OR bolus feeding

INTERVENTIONS:
Other: Method of feeding; continuous feeding OR bolus feeding — CF: Infants fed through a naso or orogastric tube in a continuous fashion using syringe pump. Each feed cycle is of 4 hours (3 hrs continuous feeding and 1 hour rest). 6 feed cycles in a day.
  BF: Infants fed through a naso or orogastric tube in a gravity dependent bolus feeding every 2-3 hours. Each feed would take approximately 10 minutes.

SUMMARY:
Chronic Lung Disease (CLD) of Prematurity is a common yet challenging co-morbidity affecting extremely premature newborns. Multifactorial influences leading to this co-morbidity is known and targeted in various research studies. Gastroesophageal reflux (GER) is common among the same cohort of patients. The investigators hypothesize that recurrent milk reflux into the airways of the premature babies worsen the inflammation of premature lungs and is a major contributor of CLD.

The investigators hypothesize that Continuous feeding (CF) minimises GER and micro-aspiration, thereby reducing the incidence and severity of CLD in high-risk infants.

Our aim is to compare the effect of intermittent bolus versus continuous intra-gastric feeding on the incidence and severity of CLD in very low birth weight infants ≤ 1250 grams.

DETAILED DESCRIPTION:
The pathogenesis of bronchopulmonary dysplasia (BPD) is complex and multifactorial. As a result of premature birth, developmental arrest during a critical period of fetal lung development compounded by mechanical, oxidative and other injuries sustained during neonatal respiratory care forms the basis of pathogenesis. BPD affects up to 50% of infants with birth weight less than 1000 g. Between 2000 and 2009, despite advancement of neonatal care, annual BPD rates reported by Vermont Oxford Network among very low birth weight infants varied from 26.2% to 30.4% without any decline. Severely affected infants often require prolonged ventilation, high oxygen use, alternative airway and several potent medications over the first few months to years of their lives. High mortality rates, neurodevelopmental delay, respiratory morbidity and growth failure are associated with BPD.

Treatment of severe BPD with or without pulmonary hypertension is challenging. Prolonging the pregnancy in the face of premature labour, treating perinatal infections, augmenting pulmonary maturity with corticosteroids, judicious oxygen use, lung protective ventilation and optimizing nutrition to promote growth are important and well established measures to prevent or modify the progress of the chronic lung disease.

It is common to find infants with BPD also having significant symptoms of reflux. Gastroesophageal reflux (GER) is a well-known co-morbidity among preterms and ex-preterms on chronic ventilation, many of whom go on to require surgical fundoplication to stop the reflux thus preventing further lung damage. Some have reported dramatic respiratory improvement after resolution of GER. In the early days of a preterm baby with respiratory distress, GER is common and silent. Among infants, diagnosis of pathologic GER from a benign one is difficult. Many neonatal intensive care units (NICUs) would investigate for GER only when faced with moderate to severe BPD to achieve better respiratory symptom control. However GER has not been studied well as a factor precipitating the development of BPD among VLBW neonates. This is the focus of the study.

Aspiration of gastric contents into the lung is a widespread phenomenon in mechanically ventilated preterm infants. In animal models of gastric aspiration, gastric particulates altered the pulmonary mechanics, increased pulmonary inflammatory cells, released pro-inflammatory mediators, and inactivated surfactant. Development of bacterial pneumonia is a well-recognized complication following aspiration of gastric contents. The investigators hypothesize that repeated aspirations would aggravate and accelerate an inflammatory response in the lung finally leading on to BPD. In addition oxygen mediated damage and mechanical ventilation potentiate lung injury due to aspiration. Logically, if GER and aspiration could be minimized, it could decrease the incidence and severity of BPD.

Certain positioning of the baby, small volume of feed increment, keeping a close watch on feed tolerance are practical ways of improving feeding tolerance and reducing GER. The intermittent bolus intra-gastric feeding method is commonly used to feed premature babies. Other alternatives are continuous intra-gastric (feed volume is slowly infused in the stomach over couple of hours through the nasogastric tube) and continuous transpyloric feeding (feeding tube passes beyond the stomach to the duodenum and feed volume is slowly infused over hours). Transpyloric continuous feeding as compared to intermittent gastric bolus feeding, has been found to significantly reduce ventilatory support requirements in extremely low birth weight (ELBW) infants, possibly via its effect of minimising GER. In this study, none of the babies who received transpyloric feeding developed significant BPD and in addition babies with significant BPD improved after switching to transpyloric method. Transpyloric feeding tubes however are challenging to insert, and intestinal perforation is an uncommon but significant adverse effect. This feeding method is also not physiological as it bypasses the stomach. It remains to be seen if continuous gastric feeds, which is easily administered and safer, would yield some of the advantages of continuous transpyloric feeds over intermittent gastric feeding.

A Cochrane review in 2011 of continuous intra-gastric versus intermittent bolus intra-gastric feeding for premature infants found conflicting results, and was unable to make recommendations regarding the benefits and risks of these feeding methods. Clinical outcomes of interest from these trials were related to growth, feeding tolerance and gastrointestinal complications. The Cochrane review importantly found no significant difference in somatic growth and incidence of necrotising enterocolitis (NEC) between either feeding methods. Another Cochrane review in 2014 did not identify any randomised trial that evaluated the effects of continuous versus intermittent bolus intragastric tube feeding on gastro-oesophageal reflux disease in preterm and low birth weight infants and opined that well-designed and adequately powered trials are needed in this field. There were no studies comparing the effect of the above feeding methods on respiratory outcomes either.

Trial objectives

Aim: To compare the effect of intermittent bolus versus continuous intra-gastric feeding on the incidence and severity of BPD in very low birth weight infants (≤ 1250 grams).

Hypothesis: Continuous feeding (CF) minimises silent GER and micro-aspiration, thereby reducing the incidence and severity of bronchopulmonary dysplasia (BPD) in high-risk infants when compared to intermittent bolus feeding (BF).

Statistical considerations

Sample size calculation: based on 2015 data from the Singapore National Very-Low-Birth-Weight (VLBW) Infant Network for infants ≤ 1250 grams, mortality rate was 12.9% and BPD rate (defined as any oxygen supplementation or any respiratory support at 36 weeks post-conceptional age) was 29.4%. Thus the composite primary outcome rate was 42.3%. For a primary outcome rate reduction from 45% to 22.5%, with a type 1 error rate of 5% and a power of 80%, a sample size of 68 infants in each arm is required, giving a total sample size of 136 infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants with a birth weight <1250g and a gestational age of between 24+0 - 33+6 weeks

Exclusion Criteria:

1. Major congenital malformation
2. Chromosomal abnormality
3. 10-minute Apgar score of =3
4. Not expected to survive beyond 72 hours of age
5. Bilateral grade 4 intraventricular haemorrhage (IVH)
6. Did not consent / Consent not available

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2019-12-03 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of BPD | occurring before 36 weeks post menstrual age or 28 days of life
  BPD as defined by 2001 NICHD criteria
Incidence of Death | occurring before 36 weeks post menstrual age or 28 days of life
  Death occurring before 36 weeks post menstrual age or 28 days of life

SECONDARY OUTCOMES:
Invasive Ventilatory requirements | 36 weeks post menstrual age or 28 days of life
  Days on invasive ventilation
Any Ventilatory requirements | 36 weeks post menstrual age or 28 days of life
  Days on any ventilatory (invasive or non invasive) support
Supplemental Oxygen support | 36 weeks post menstrual age or 28 days of life
  Days on supplemental oxygen
Feed tolerance | 36 weeks post menstrual age or 28 days of life
  Time (days) from randomization to achievement of full feeds (defined as 150ml/Kg/Day)
Weight outcomes | birth, 36 weeks and 40 weeks post menstrual age
  Z-scores for weight (grams)
Length outcomes | birth, 36 weeks and 40 weeks post menstrual age
  Z-scores for length (cm)
Head Growth outcomes | birth, 36 weeks and 40 weeks post menstrual age
  Z-scores for head circumference (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Agnihotri Biswas, MRCPCH, Principal Investigator — Senior Consultant Neonatologist, NUH Singapore
Locations (2):
- NICU, Universiti Kebangsaan Malaysia, Kuala Lumpur, Malaysia
- NICU, National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bancalari E, Claure N, Sosenko IR. Bronchopulmonary dysplasia: changes in pathogenesis, epidemiology and definition. Semin Neonatol. 2003 Feb;8(1):63-71. doi: 10.1016/s1084-2756(02)00192-6. PMID 12667831
- [Background] Stoll BJ, Hansen NI, Bell EF, Shankaran S, Laptook AR, Walsh MC, Hale EC, Newman NS, Schibler K, Carlo WA, Kennedy KA, Poindexter BB, Finer NN, Ehrenkranz RA, Duara S, Sanchez PJ, O'Shea TM, Goldberg RN, Van Meurs KP, Faix RG, Phelps DL, Frantz ID 3rd, Watterberg KL, Saha S, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Neonatal outcomes of extremely preterm infants from the NICHD Neonatal Research Network. Pediatrics. 2010 Sep;126(3):443-56. doi: 10.1542/peds.2009-2959. Epub 2010 Aug 23. PMID 20732945
- [Background] Horbar JD, Carpenter JH, Badger GJ, Kenny MJ, Soll RF, Morrow KA, Buzas JS. Mortality and neonatal morbidity among infants 501 to 1500 grams from 2000 to 2009. Pediatrics. 2012 Jun;129(6):1019-26. doi: 10.1542/peds.2011-3028. Epub 2012 May 21. PMID 22614775
- [Background] Ehrenkranz RA, Walsh MC, Vohr BR, Jobe AH, Wright LL, Fanaroff AA, Wrage LA, Poole K; National Institutes of Child Health and Human Development Neonatal Research Network. Validation of the National Institutes of Health consensus definition of bronchopulmonary dysplasia. Pediatrics. 2005 Dec;116(6):1353-60. doi: 10.1542/peds.2005-0249. PMID 16322158
- [Background] Jobe AH. The new bronchopulmonary dysplasia. Curr Opin Pediatr. 2011 Apr;23(2):167-72. doi: 10.1097/MOP.0b013e3283423e6b. PMID 21169836
- [Background] Cristea AI, Carroll AE, Davis SD, Swigonski NL, Ackerman VL. Outcomes of children with severe bronchopulmonary dysplasia who were ventilator dependent at home. Pediatrics. 2013 Sep;132(3):e727-34. doi: 10.1542/peds.2012-2990. Epub 2013 Aug 5. PMID 23918888
- [Background] Walsh MC, Morris BH, Wrage LA, Vohr BR, Poole WK, Tyson JE, Wright LL, Ehrenkranz RA, Stoll BJ, Fanaroff AA; National Institutes of Child Health and Human Development Neonatal Research Network. Extremely low birthweight neonates with protracted ventilation: mortality and 18-month neurodevelopmental outcomes. J Pediatr. 2005 Jun;146(6):798-804. doi: 10.1016/j.jpeds.2005.01.047. PMID 15973322
- [Background] Khemani E, McElhinney DB, Rhein L, Andrade O, Lacro RV, Thomas KC, Mullen MP. Pulmonary artery hypertension in formerly premature infants with bronchopulmonary dysplasia: clinical features and outcomes in the surfactant era. Pediatrics. 2007 Dec;120(6):1260-9. doi: 10.1542/peds.2007-0971. PMID 18055675
- [Background] Radford PJ, Stillwell PC, Blue B, Hertel G. Aspiration complicating bronchopulmonary dysplasia. Chest. 1995 Jan;107(1):185-8. doi: 10.1378/chest.107.1.185. PMID 7813274
- [Background] Demirel G, Yilmaz Y, Uras N, Erdeve O, Ulu HO, Oguz SS, Dilmen U. Dramatical recovery of a mechanical ventilatory dependent extremely low birth weight premature infant after Nissen fundoplication. J Trop Pediatr. 2011 Dec;57(6):484-6. doi: 10.1093/tropej/fmq125. Epub 2011 Jan 19. PMID 21252395
- [Background] Gien J, Kinsella J, Thrasher J, Grenolds A, Abman SH, Baker CD. Retrospective Analysis of an Interdisciplinary Ventilator Care Program Intervention on Survival of Infants with Ventilator-Dependent Bronchopulmonary Dysplasia. Am J Perinatol. 2017 Jan;34(2):155-163. doi: 10.1055/s-0036-1584897. Epub 2016 Jun 29. PMID 27355979
- [Background] Newell SJ, Booth IW, Morgan ME, Durbin GM, McNeish AS. Gastro-oesophageal reflux in preterm infants. Arch Dis Child. 1989 Jun;64(6):780-6. doi: 10.1136/adc.64.6.780. PMID 2774613
- [Background] Ewer AK, Durbin GM, Morgan ME, Booth IW. Gastric emptying and gastro-oesophageal reflux in preterm infants. Arch Dis Child Fetal Neonatal Ed. 1996 Sep;75(2):F117-21. doi: 10.1136/fn.75.2.f117. PMID 8949695
- [Background] Peter CS, Sprodowski N, Bohnhorst B, Silny J, Poets CF. Gastroesophageal reflux and apnea of prematurity: no temporal relationship. Pediatrics. 2002 Jan;109(1):8-11. doi: 10.1542/peds.109.1.8. PMID 11773535
- [Background] Lopez-Alonso M, Moya MJ, Cabo JA, Ribas J, del Carmen Macias M, Silny J, Sifrim D. Twenty-four-hour esophageal impedance-pH monitoring in healthy preterm neonates: rate and characteristics of acid, weakly acidic, and weakly alkaline gastroesophageal reflux. Pediatrics. 2006 Aug;118(2):e299-308. doi: 10.1542/peds.2005-3140. Epub 2006 Jul 10. PMID 16831894
- [Background] Fuloria M, Hiatt D, Dillard RG, O'Shea TM. Gastroesophageal reflux in very low birth weight infants: association with chronic lung disease and outcomes through 1 year of age. J Perinatol. 2000 Jun;20(4):235-9. doi: 10.1038/sj.jp.7200352. PMID 10879336
- [Background] Jadcherla SR, Peng J, Chan CY, Moore R, Wei L, Fernandez S, DI Lorenzo C. Significance of gastroesophageal refluxate in relation to physical, chemical, and spatiotemporal characteristics in symptomatic intensive care unit neonates. Pediatr Res. 2011 Aug;70(2):192-8. doi: 10.1203/PDR.0b013e31821f704d. PMID 21730816
- [Background] Farhath S, He Z, Nakhla T, Saslow J, Soundar S, Camacho J, Stahl G, Shaffer S, Mehta DI, Aghai ZH. Pepsin, a marker of gastric contents, is increased in tracheal aspirates from preterm infants who develop bronchopulmonary dysplasia. Pediatrics. 2008 Feb;121(2):e253-9. doi: 10.1542/peds.2007-0056. PMID 18245400
- [Background] Knight PR, Davidson BA, Nader ND, Helinski JD, Marschke CJ, Russo TA, Hutson AD, Notter RH, Holm BA. Progressive, severe lung injury secondary to the interaction of insults in gastric aspiration. Exp Lung Res. 2004 Oct-Nov;30(7):535-57. doi: 10.1080/01902140490489162. PMID 15371091
- [Background] Davidson BA, Knight PR, Wang Z, Chess PR, Holm BA, Russo TA, Hutson A, Notter RH. Surfactant alterations in acute inflammatory lung injury from aspiration of acid and gastric particulates. Am J Physiol Lung Cell Mol Physiol. 2005 Apr;288(4):L699-708. doi: 10.1152/ajplung.00229.2004. PMID 15757954
- [Background] Nader-Djalal N, Knight PR, Davidson BA, Johnson K. Hyperoxia exacerbates microvascular lung injury following acid aspiration. Chest. 1997 Dec;112(6):1607-14. doi: 10.1378/chest.112.6.1607. PMID 9404761
- [Background] Nader-Djalal N, Knight PR 3rd, Thusu K, Davidson BA, Holm BA, Johnson KJ, Dandona P. Reactive oxygen species contribute to oxygen-related lung injury after acid aspiration. Anesth Analg. 1998 Jul;87(1):127-33. doi: 10.1097/00000539-199807000-00028. PMID 9661561
- [Background] Hermon MM, Wassermann E, Pfeiler C, Pollak A, Redl H, Strohmaier W. Early mechanical ventilation is deleterious after aspiration-induced lung injury in rabbits. Shock. 2005 Jan;23(1):59-64. doi: 10.1097/01.shk.0000143417.28273.6d. PMID 15614133
- [Background] Premji SS, Chessell L. Continuous nasogastric milk feeding versus intermittent bolus milk feeding for premature infants less than 1500 grams. Cochrane Database Syst Rev. 2011 Nov 9;2011(11):CD001819. doi: 10.1002/14651858.CD001819.pub2. PMID 22071802
- [Background] Richards R, Foster JP, Psaila K. Continuous versus bolus intragastric tube feeding for preterm and low birth weight infants with gastro-oesophageal reflux disease. Cochrane Database Syst Rev. 2014 Jul 17;(7):CD009719. doi: 10.1002/14651858.CD009719.pub2. PMID 25030383
- [Background] de Ville K, Knapp E, Al-Tawil Y, Berseth CL. Slow infusion feedings enhance duodenal motor responses and gastric emptying in preterm infants. Am J Clin Nutr. 1998 Jul;68(1):103-8. doi: 10.1093/ajcn/68.1.103. PMID 9665103
- [Background] Jobe AH, Bancalari E. Bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2001 Jun;163(7):1723-9. doi: 10.1164/ajrccm.163.7.2011060. No abstract available. PMID 11401896